CLINICAL TRIAL: NCT03768986
Title: A Reinforcement Intervention for Increasing HIV Testing Among At-Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Kristyn Zajac, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-018-1; R01MD013550 (NIH)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: HIV; HIV Testing; Women; Contingency Management
MeSH Terms: interventions — HIV Testing; Reinforcement Machine Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group A (Active Comparator): Standard referral for HIV testing and online HIV risk reduction training
  Interventions: Behavioral: Standard referral for HIV testing; Behavioral: Online risk reduction training
- Treatment Group B (Experimental): Standard referral for HIV testing and online HIV risk reduction training plus reinforcement
  Interventions: Behavioral: Standard referral for HIV testing; Behavioral: Online risk reduction training; Behavioral: Reinforcement

INTERVENTIONS:
Behavioral: Standard referral for HIV testing — Participants receive standard referral for HIV testing in the community.
Behavioral: Online risk reduction training — Participants are encouraged to use the CDC's website to learn more about their individual risks for HIV and how to reduce them.
Behavioral: Reinforcement — Systematic reinforcement of desired behaviors Participants will receive a monetary incentive for getting tested for HIV
  Arms: Treatment Group B

SUMMARY:
African American and Latina women, as well as women living in poverty, are an identified health disparities population for HIV. Risks for HIV are compounded in this population when additional risk factors are present, including other sexually transmitted infections, intimate partner violence, substance use disorders, and homelessness or housing insecurity. Knowledge of one's HIV serostatus is key to linkage to care, improving HIV outcomes, and decreasing the spread of HIV. However, roughly a third of African American women and over half of Latina women have never been tested (CDC, 2016a). Barriers to testing include socioeconomical inequality, racial discrimination, low health literacy, and inadequate access to quality healthcare, among others. Novel methods for increasing HIV testing in this important health disparities group are greatly needed.

This study aims to test a reinforcement-based intervention to increase HIV testing and repeat testing among African American, Latina, and women living in poverty who have risk factors for HIV. We are partnering with multiple community-based organizations, several of which are non-traditional providers of HIV services (e.g., domestic violence agency, homeless shelter), to address systemic and structural issues that serve as barriers to testing. A primary aim is to evaluate the effectiveness of training community-based providers to deliver a reinforcement-based intervention for promoting HIV testing. In addition, we will compare standard referral services for HIV testing plus HIV risk reduction education to the same plus reinforcement for HIV testing (and repeat testing) using a randomized controlled trial with 334 participants. Women in both groups will be encouraged to seek HIV testing; be provided with the resources to do so (list of testing sites, bus passes if needed); and will receive basic education about HIV prevention using a widely available web-based resource (https://wwwn.cdc.gov/hivrisk/). Women in the reinforcement group will also be provided with $25 for undergoing an HIV test, with a $15 bonus if they have the test in the next 7 days ($40 total). During the next 12 months, they can receive an additional $25 for undergoing up to 2 more tests separated by 12 weeks, with $15 bonuses for each test completed within 7 days (+/- 7 days) of the scheduled date at 6- and 12-months post-initial test. It is hypothesized that the reinforcement intervention will result in greater proportions of women receiving an HIV test (and repeat HIV tests) compared to standard services.

In the proposed study, approximately 50 clinicians from our partner sites will be trained on both the non-reinforcement and reinforcement approaches to increasing HIV testing. Primary clinician outcomes are clinician knowledge and attitudes about HIV, testing, and reinforcement interventions. These will be assessed pre- and post-training and at 6-month intervals thereafter. A secondary outcome is clinician satisfaction with the training. Once clinicians are trained to competence, 334 women at our partner agencies will be randomized. Participants will be assessed at baseline and at 3-, 9-, and 15-month follow-ups. The primary outcome is objective reports of HIV testing, verified by testing centers. Secondary outcomes are HIV risk behaviors, test results, self-efficacy, client attitudes towards testing, and HIV knowledge. In addition, this study will include a careful analysis of costs of the reinforcement intervention to allow for estimates of its cost-effectiveness in increasing HIV testing.

The overall goal of this study is to determine whether a reinforcement intervention delivered by community providers is superior to standard referral procedures plus HIV education in increasing rates of HIV testing among women at the highest risk of HIV infection. A wide range of community partners that serve some of the highest risk groups of women were chosen to ensure highly generalizable results. If efficacious, the intervention has the potential for widespread adoption and implementation.

ELIGIBILITY:
Inclusion Criteria for Clinician Participants:

* >6 months experience as a case manager, medical/nursing clinician or mental health/substance use therapist
* currently work with women at high risk for contracting HIV
* able to attend a training and participate in the evaluative components
* willing to conduct both standard HIV referral for testing and orientation to an online training and the same with reinforcement, depending on client's random assignment.

Exclusion Criteria for Clinician Participants

- planning to end employment at the agency within the next 3 months

Inclusion Criteria for Client Participants:

* female
* identifies as African American/black or Latina/Hispanic OR is living in poverty based on the most recent year's federal poverty guidelines
* 18 and older
* one or more high risk factors for HIV: intravenous drug use; or sexually active with past year partners with HIV or of unknown HIV status and no or inconsistent use of condoms
* English or Spanish speaking
* passes a quiz related to understanding the informed consent form
* has an address at which they expect to be able to receive mail and/or a phone to retrieve messages for the next 15 months

Exclusion Criteria for Client Participants:

* received a fourth-generation HIV test in the past 6 months
* HIV positive.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
HIV testing by clients | From date of intervention until date of documented HIV test, assessed up to 15 months
  HIV testing completion (i.e. having test completed) will be verified by the testing sites
Clinician knowledge | Baseline and immediately post-training
  Change in clinician knowledge will be measured through self-reports

SECONDARY OUTCOMES:
Clinician satisfaction with training | Post-training, up to 1 month
  Satisfaction with training will be measured by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Zajac, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No